CLINICAL TRIAL: NCT06420336
Title: Quadratus Lumborum Block for Pain Control in Unilateral Anterior Iliac Bone Graft Harvesting for Pediatric Patients Undergoing Palatoplasty: a Prospective Randomized Control Trial
Brief Title: QL vs LAI for Palatoplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Nicole McCoy, Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00136697
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Post-operative Pain; Opioid Use; Cleft Palate
MeSH Terms: conditions — Pain, Postoperative; Cleft Palate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quadratus lumborum block (Active Comparator): After induction of anesthesia and securement of appropriate airway device, the patient will be placed in position for the QL block. Using ultrasound guidance, the pediatric anesthesiology attending will perform unilateral QL block on the side of the anterior iliac bone graft harvest. The dose will be 0.2% ropivacaine, 1 mL per kilogram to a max of 20 mL with an additive of dexamethasone 4 mg. Ultrasonography will be used to identify external oblique, internal oblique, transverse abdominus and quadratus lumborum muscles. A 50 mm-150 mm block needle will be advanced under ultrasound guidance. Ropivacaine will be injected slowly with frequent aspiration to rule out incorrect needle placement. The anesthetic is deposited at the lateral edge of the QL after penetrating the transversus abdominus aponeurosis. Injection will continue to be observed with real time US guidance.
  Interventions: Procedure: Quadratus lumborum block
- Local anesthetic infiltration (Active Comparator): Patient will undergo induction of anesthesia as deemed appropriate by the attending pediatric anesthesiologist assigned to the case. After induction of anesthesia and securement of appropriate airway device the patient will be turned over to the surgical team to proceed with the operation. The surgeon will proceed with usual injection of local anesthetic as their standard of care; this medication will be charted by the circulating nurse in the Medication Administration Record with local anesthetic type and amount. At the conclusion of the procedure, to maintain the blind, the patient will have a bandage placed where the QL block would have been performed.
  Interventions: Procedure: Local anesthetic infiltration

INTERVENTIONS:
Procedure: Quadratus lumborum block — After induction of anesthesia and securement of appropriate airway device, the patient will be placed in position for the QL block. Using ultrasound guidance, the pediatric anesthesiology attending will perform unilateral QL block on the side of the anterior iliac bone graft harvest. The dose will be 0.2% ropivacaine, 1 mL per kilogram to a max of 20 mL with an additive of dexamethasone 4 mg. Ultrasonography will be used to identify external oblique, internal oblique, transverse abdominus and quadratus lumborum muscles. A 50 mm-150 mm block needle will be advanced under ultrasound guidance. Ropivacaine will be injected slowly with frequent aspiration to rule out incorrect needle placement. The anesthetic is deposited at the lateral edge of the QL after penetrating the transversus abdominus aponeurosis. Injection will continue to be observed with real time US guidance.
  Arms: Quadratus lumborum block
Procedure: Local anesthetic infiltration — After induction of anesthesia and securement of appropriate airway device the patient will be turned over to the surgical team to proceed with the operation. The surgeon will proceed with usual injection of local anesthetic as their standard of care; this medication will be charted by the circulating nurse in the Medication Administration Record with local anesthetic type and amount. At the conclusion of the procedure, to maintain the blind, the patient will have a bandage placed where the QL block would have been performed.
  Arms: Local anesthetic infiltration

SUMMARY:
This study will consist of patients ages 6-18 who are undergoing a surgery on the hard or soft palate of the mouth (palatoplasty), with removal of bone from the front of the hip (anterior iliac bone graft harvesting). The patients will be randomized to receive either a unilateral QL block by an anesthesiologist, or local anesthetic infiltration at the surgical incision by the surgeon. The primary aim will be assessing post-operative pain in the first 48 hours after surgery. Secondary outcomes will include pain medication use in the first 48 hours after surgery, block resolution time, and evaluating any complications associated with the QL block or local anesthetic infiltration.

ELIGIBILITY:
Inclusion Criteria

* Patients undergoing palatoplasty with autologous bone graft from the anterior iliac crest.
* Ages 6-18 years of age
* Planned admission post-op
* ASA Status Range: 1-3

Exclusion Criteria

* Contraindication to QL blocks or LAI which may include:
* overlying infection skin at the block needle insertion site
* coagulopathies
* known bleeding disorders
* Allergy to local anesthetic
* Cognitive or developmental impairment that would limit ability to report pain.
* Non-English Speaking/Writing
* Subjects or their parent/guardian unable or choose to not give informed consent/assent.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | 0-48 hours after surgery ends
  Using the Wong-Baker FACES Pain Rating Scale, patients will report their average pain from 0 hours post-op through 48-hours post-op at various intervals. In the Post-Anesthesia Recovery Unit, pain scores will be evaluated every 15 minutes as clinically able, until discharged from the PACU. On Post-Op Day 1 at 9:00 am, pains average pain score from discharge to PACU to midnight will be reported. At approximately 24-hours after surgery ends, pain scores from midnight to 23-hours post-op will be reported, then at the 48-hour post-op mark, pain scores from 24-hr post op to 48-hour post-op time will be recorded.

SECONDARY OUTCOMES:
Time to block resolution | up to 7 days after surgery ends
  Subjects will report the date and time that resolution of numbness over operative hip occurs or feeling of pain in operative hip returns.
Opioid Consumption up to 48 hours after surgery ends | From the pre-operative phase up to 48 hours after surgery ends
  Total morphine milligram equivalents (MME) will be calculated from pre-op to 48-hours after surgery ends.
Number of complications associated with each intervention | From the time the intervention is administered up to 48-hours after surgery ends.
  Complications associated with study participation will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole McCoy, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No